CLINICAL TRIAL: NCT06132776
Title: High Tone Therapy for Chemotherapy-induced Neuropathy in Breast Cancer Patients
Brief Title: The Mamma HiToP Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Hospital Association (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP_Mamma 1.1
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum group (Experimental)
  Interventions: Device: HiToP 191 PNP
- Placebo group (Placebo Comparator)
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: HiToP 191 PNP — High tone therapy
  Arms: Verum group
Device: Placebo device — Placebo therapy
  Arms: Placebo group

SUMMARY:
The HiToP ® 191 PNP an certified device licensed for the treatment of neuropathia.

The home-based treatment is to be performed only in accordance with the approved Investigational Plan (CIP) on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

The study is multicenter, randomized, double-blind, and placebo-controlled.

Primary Objective: Comparison of the change of paresthesias from baseline until end of therapy between the two patient groups, assessed by questionnaires

Secondary Objectives: Further symptoms of neuropathy as well as on health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with histologically verified breast cancer and neoadjuvant or adjuvant treatment with a taxane derivate (e.g., Paclitaxel, Docetaxel): This group was chosen due to relatively high risk of neuropathy due to this special therapeutic agent 1,9.
* Cumulative dose of at least 3 cycles
* Interval of 2 weeks since the last chemotherapeutic cycle in order to prevent false worsenings due to delayed neurotoxic effects
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2 (that is, the capability to walk and to spend less than 50% of waking hours sitting or lying)
* Ability to walk (with or without aids)
* European Organisation for Research and Treatment of Cancer (EORTC) common toxicity criteria (CTC) peripheral sensory neuropathy grade 1 or 2
* Intensity of paresthesias of > 3/10 on the Visual Analog Scale (VAS)

Exclusion Criteria:

* - Prevalent neuropathy of different etiology
* Serious central-neurological or psychiatric disorder that would interfer with a proper order of the study, according to the judgement of the investigators
* Epilepsy
* Minors or persons unable to give informed consent
* Current neurotoxic medication
* Implanted pacemakers or defibrillators
* Pregnancy
* Wounds in the area to be treated, acute local or systemic infection
* Peripheral arterial occlusive disease > grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Alleviation of paresthesias (VAS) | baseline vs. one day after the last treatment session
  Visual analog scale, 0-10, higher score = worse

SECONDARY OUTCOMES:
Further neuropathic symptoms (via VAS questionnaire) | baseline vs. one day after the last treatment session vs. follow-up 2 weeks after the last treatment session
  e.g., intensity of tightness, cramps, 0-10, higher score = worse
Further neuropathic symptoms (via EORCT CIPN20 questionnaire) | baseline vs. one day after the last treatment session vs. follow-up 2 weeks after the last treatment session
  sensory, motor and autonomic scale, 1-4, higher score = worse
Quality of life (via EORCT C30 questionnaire) | baseline vs. one day after the last treatment session vs. follow-up 2 weeks after the last treatment session
  global health status, physical function, symptom scales, 1-4, higher score = worse

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Paternostro-Sluga, MD, Study Director — Vienna Healthcare Group
Locations (1):
- Clinics Donaustadt, Ottakring, Hietzing, Vienna, Austria